CLINICAL TRIAL: NCT03418129
Title: Neuromodulatory Treatments for Pain Management in Veterans With Complex TBI Using Mobile Technology
Brief Title: Neuromodulatory Treatments for Pain Management in TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00088360
Record Dates: First submitted 2017-11-03; First posted 2018-02-01 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pain; Traumatic Brain Injury; Posttraumatic Stress Disorder
Keywords: Military Veterans
MeSH Terms: conditions — Chronic Pain; Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Mobile App Mindfulness (Experimental): Participants engage in the use of a mobile application on an iPod Touch for a minimum of 10 minutes a day, 4 days a week for a total of 12 weeks.
  Interventions: Device: Mindfulness
- Mobile App Neurofeedback (Experimental): Participants engage in use of a mobile application on an iPod Touch for a minimum of 10 minutes a day, 4 days a week for a total of 12 weeks.
  Interventions: Device: Neurofeedback
- Mobile App Relaxation (Experimental): Participants engage in use of a mobile application on an iPod Touch for a minimum of 10 minutes a day, 4 days a week for a total of 12 weeks.
  Interventions: Device: Relaxation

INTERVENTIONS:
Device: Mindfulness — Neuromodulatory intervention for pain management
  Arms: Mobile App Mindfulness
Device: Neurofeedback — Neuromodulatory intervention for pain management
  Arms: Mobile App Neurofeedback
Device: Relaxation — Neuromodulatory intervention for pain management
  Arms: Mobile App Relaxation

SUMMARY:
Traumatic brain injury (TBI) and chronic pain are common and serious health problems for military veterans and often co-occur, leading to poor post-deployment adjustment. Pharmacological treatments for pain elevate risk of opioid abuse, and research suggests veterans perceive barriers to existing non-pharmacological, clinic-based treatments. Thus, there is an urgent need to develop pain management approaches that are effective, overcome barriers to care, and are readily usable by Veterans. Evidence suggests that neuromodulatory treatments, grounded in understanding of neurophysiological mechanisms of pain, reduce pain-related symptoms and have the potential to be developed into self-directed treatments through use of mobile technology.

DETAILED DESCRIPTION:
This study is a prospective, three-arm, randomized controlled trial of neuromodulatory treatments for chronic pain, for post-9/11 veterans with co-occuring pain and TBI. Three hundred participants will be scheduled for a baseline interview at the Duke Behavioral Health and Technology Lab after passing a preliminary telephone screen. After providing informed consent, participants will provide data on clinical measures. Electroencephalography (EEG) will be used to measure brain activity. Following data collection, participants will be assigned to one of three groups (n=100 in each). Each group will receive an iPod Touch with a different mobile application (app), which participants will be instructed to use for 10 minute a day, 4 times a week for 12 weeks. Study coordinators will conduct two home visits (week 1 and week 6) and two phone calls (week 3 and week 9) to reinforce training, troubleshoot difficulties, and ask about intervention utilization. Follow-up data on clinical measures and EEG will be collected at 12 weeks and again at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Served in one of the military branches (Army, Navy, Marines, Air Force, or Coast Guard) since October 2001.
2. Diagnosis of Traumatic Brain Injury (TBI), defined as a traumatically induced structural injury or physiological disruption of brain function, as a result of an external force, that is indicated by new or onset or worsening of at least one of the following signs immediately following the event:

   * Any alteration in mental status (e.g. confusion, disorientation, slowed thinking, etc.)
   * Any loss of memory for events immediately before or after the injury.
   * Any period of loss or a decreased level of consciousness, observed or self-reported.
3. Reports chronic musculoskeletal and/or neuropathic pain, defined as moderate or severe pain (≥ 4 on a 0-10 rating scale) in one or more body regions for the previous 3 months or more. For individuals on pain medication, inclusion criteria are that (a) their pain medication regimen has been stable for the past 4 weeks, (b) they do not expect any major changes in their pain medication regimen for the duration of the study, and (c) they do not expect to have surgery or to be hospitalized for pain treatment for the duration of the study.

Exclusion Criteria:

1. History of epilepsy, seizure disorder, or any seizure or epileptic fit.
2. Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Elbogen, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Department of Psychiatry, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Per FITBIR (Federal Interagency Traumatic Brain Injury Research) policy on Data Sharing, we will submit all de-identified data to FITBIR after the completion of the study. All data are submitted in accord with applicable laws and regulations, and that the identities of research participants will not be disclosed to the FITBIR Informatics System. FITBIR Data Sharing Policy includes steps to protect the interests and privacy concerns of individuals, families, and identifiable groups who participate in TBI genetic and other research.
Time Frame: A contribution will be submitted after study completion and will remain in the FITBIR database indefinitely.
Access Criteria: Only individuals with a FITBIR account who have submitted a Data Access Request that has been reviewed by the Data Access Quality Committee will be able to view the data.
URL: https://fitbir.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile App Mindfulness | Mobile App Neurofeedback | Mobile App Relaxation
Started | 84 | 85 | 85
Completed | 70 | 59 | 66
Not Completed | 14 | 26 | 19
Not completed — Lost to Follow-up | 11 | 20 | 15
Not completed — Withdrawal by Subject | 3 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile App Mindfulness | Mobile App Neurofeedback | Mobile App Relaxation | Total
Number analyzed (Participants) | 84 | 85 | 85 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.45 (8.78) | 41.99 (9.27) | 40.69 (8.63) | 41.38 (8.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 20 | 17 | 50
  Male | 71 | 65 | 68 | 204
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 12 | 7 | 25
  Not Hispanic or Latino | 70 | 65 | 61 | 196
  Unknown or Not Reported | 8 | 8 | 17 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5 | 10
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 3 | 5
  Black or African American | 14 | 13 | 13 | 40
  White | 63 | 65 | 58 | 186
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 6 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 84 | 85 | 85 | 254

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-reported Pain Intensity
Description: Measured by the Defense and Veterans Pain Rating Scale (DVPRS), a graphic tool to facilitate self-reported pain rating using a scale from 0-10, 0 being "no pain" to 10 being "as bad as it could be, nothing else matters."
Time Frame: Baseline and 12 weeks
Population: Participants who completed the DVPRS at 0 and 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile App Mindfulness | Mobile App Neurofeedback | Mobile App Relaxation
Number analyzed (Participants) | 75 | 68 | 76
score on a scale | -1.02 (1.32) | -0.78 (1.27) | -1.03 (1.36)
Statistical Analysis 1: Comparison: Mobile App Neurofeedback vs Mobile App Relaxation; Test type: Superiority; p = 0.2852, ANCOVA; Slope = 0.2331, Standard Error of Mean 0.2176 — Multilevel modeling was used to model outcome at baseline and 3-month follow-up. Resulting slopes capture change in outcome from baseline to follow-up, with relaxation set as the comparison
Statistical Analysis 2: Comparison: Mobile App Mindfulness vs Mobile App Relaxation; Test type: Superiority; p = 0.8861, ANCOVA; Slope = 0.03057, Standard Error of Mean 0.2132 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change in EEG Alpha Power
Description: Average FFT (Fast Fourier Transform) Power (alpha 8-12 Hz) measured as sqrt(uV)/Hz.
Time Frame: 0 and 12 weeks
Population: EEG measurement was discontinued in March 2020 due to the COVID pandemic. Data not collected on 127 participants.
Measure: Mean (Standard Deviation); unit: sqrt(uV)/Hz
Arm/Group | Mobile App Mindfulness | Mobile App Neurofeedback | Mobile App Relaxation
Number analyzed (Participants) | 41 | 43 | 43
sqrt(uV)/Hz | -0.21 (0.40) | -0.1 (0.41) | -0.07 (0.35)
Statistical Analysis 1: Comparison: Mobile App Neurofeedback vs Mobile App Relaxation; Test type: Superiority; p = 0.6842, ANOVA; Slope = -0.03844, Standard Error of Mean 0.09424 — Multilevel modeling was used to model outcomes at two time points (3-month follow-up and baseline) and across three treatment groups (Mindfulness, Neurofeedback, and Relaxation)
Statistical Analysis 2: Comparison: Mobile App Mindfulness vs Mobile App Relaxation; Test type: Superiority; p = 0.132, ANOVA; Slope = -0.1432, Standard Error of Mean 0.09427 — [estimate comment as in outcome 2, analysis 1]

3. Other Pre Specified Outcome: Change in Self-reported Pain Intensity
Description: Measured by the Defense and Veterans Pain Rating Scale (DVPRS), a graphic tool to facilitate self-reported pain rating using a scale from 0-10, 0 being "no pain" to 10 being "as bad as it could be, nothing else matters." This mean difference represents the mean change in pain intensity between 0 and 24 weeks. Please note that the analysis of results utilized a multilevel modeling (MLM) approach of all available data, which involved analyzing pain intensity data collected at 0, 12, and 24 weeks.
Time Frame: Baseline and 24 weeks
Population: Participants who completed the DVPRS at baseline, 12 weeks, and 24 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile App Mindfulness | Mobile App Neurofeedback | Mobile App Relaxation
Number analyzed (Participants) | 71 | 58 | 63
score on a scale | -1.22 (1.73) | -0.98 (1.36) | -0.86 (1.56)
Statistical Analysis 1: Comparison: Mobile App Neurofeedback vs Mobile App Relaxation; Test type: Superiority; p = 0.4542, ANCOVA; Slope = 0.1911, Standard Error of Mean 0.2551
Statistical Analysis 2: Comparison: Mobile App Mindfulness vs Mobile App Relaxation; Test type: Superiority; p = 0.1261, ANCOVA; Slope = -0.3761, Standard Error of Mean 0.2454

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Mobile App Mindfulness | Mobile App Neurofeedback | Mobile App Relaxation
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/85 | 0/85
Serious Adverse Events (participants affected / at risk) | 5/84 | 5/85 | 3/85
Other Adverse Events (participants affected / at risk) | 24/84 | 27/85 | 36/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mobile App Mindfulness (N=84) | Mobile App Neurofeedback (N=85) | Mobile App Relaxation (N=85)
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0 — Unrelated to study.
Anxiety (General disorders) | 1 | 0 | 1 — Unrelated to study.
Dizziness (General disorders) | 1 | 0 | 0 — Unrelated to study.
Headaches (General disorders) | 2 | 3 | 1 — Unrelated to study.
Blood Clot (Blood and lymphatic system disorders) | 0 | 1 | 0 — Unrelated to study.
Hospitalization (General disorders) | 0 | 1 | 1 — Unrelated to study.
Suicidality (General disorders) | 0 | 1 | 0 — Unrelated to study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mobile App Mindfulness (N=84) | Mobile App Neurofeedback (N=85) | Mobile App Relaxation (N=85)
Drowsiness (General disorders) | 20 | 17 | 16
Irritability (General disorders) | 2 | 13 | 13
Suicidal Ideation (General disorders) | 2 | 1 | 9 — Unrelated to study.

LIMITATIONS AND CAVEATS:
Due to the COVID pandemic, EEG measurement was discontinued March 2020. As a result, although all available data are provided, less than half the sample had EEG data collected and therefore analyses of this outcome measure were not powered according to original power estimates. Consequently, there can be very limited interpretation of this data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT03418129/Prot_SAP_000.pdf